CLINICAL TRIAL: NCT03308734
Title: Effects of 6 Week Reduced Exertion High Intensity Interval Training Protocol in Patients With Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resource from collaborating organisation
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, James Turner, Ph.D., FHEA, Principal Investigator, Lecturer in Human Physiology, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Prostate REHIT
Record Dates: First submitted 2017-10-01; First posted 2017-10-13 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
Keywords: High-intensity interval training; REHIT; Prostate cancer; cardiorespiratory fitness
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention Group (Experimental): Reduced-Exertion High-Intensity Interval Training Following baseline testing, participants will start a 6-week training protocol involving reduced-exertion high-intensity training on a cycle ergometer based in a gym in Gloucestershire used by the Macmillan Cancer Support's Next Steps project.
  Interventions: Behavioral: Reduced-Exertion High-Intensity Interval Training
- Control Group (No Intervention): Following baseline testing, participants will receive usual care only.

INTERVENTIONS:
Behavioral: Reduced-Exertion High-Intensity Interval Training — The 6-week REHIT protocol will involve 3 training sessions a week. Each session will include 10 minutes of unloaded pedalling using a cycle ergometer. Volunteers will be asked to increase to their maximal pedal frequency possible for 1-2 seconds prior to applying a resistance of 5 % of pre-training body weight for the Wingate sprint. The sprints will take place at 2 minutes and at 6 minutes. Sprint duration will be increased from 10 seconds in the first week to 15 seconds in the second and third weeks and finally 20 seconds in the remaining weeks. Patients will receive strong verbal encouragement during the sprints after which the resistance will be removed.
  Other Names: REHIT
  Arms: Exercise Intervention Group

SUMMARY:
Prostate cancer is the cause of the greatest number of years lived with disability due to cancer. Treatment for prostate cancer is associated with significant side effects, such as fatigue, loss of muscle mass, strength and reduced quality of life. Cardiovascular disease risk is also increased and accounts for the largest cause of mortality in these patients.

Exercise and physical activity are known to have benefits in patients with prostate cancer but time, motivation and enjoyment are often barriers. Reduced Exertion High-Intensity Interval Training (REHIT) interventions in the general population achieve similar or greater physiological benefits to continuous moderate intensity exercise but for less time commitment. Higher intensity training is also perceived as more enjoyable in both healthy populations and cancer survivors. REHIT could therefore be a potential solution to these barriers.

The aim of this project is to investigate whether a REHIT intervention results in improved cardiorespiratory fitness in patients with prostate cancer. 30 patients will be recruited and randomised to a control group or the intervention group. Both groups will undergo cardiorespiratory fitness testing pre- and post- the 6 week period of the trial. The intervention group will take part in REHIT using maximal oxygen uptake capacity (VO2 MAX) measured on a cycle ergometer. The REHIT intervention will be over 6 weeks, involving 3 sessions per week lasting 10 min and incorporating 2 Wingate sprints of 20 seconds. Pre-intervention values for VO2MAX will be compared to post-intervention values to establish whether REHIT improves cardiorespiratory function in patients with prostate cancer.

DETAILED DESCRIPTION:
Background

Among all cancers, the diagnosis of prostate cancer is associated with the greatest number of years lived with the disability and side effects of cancer. The treatment of men with prostate cancer can have a significant adverse effect on physical health. One of the primary treatment modalities is androgen-deprivation therapy which can be associated with reduced muscle mass, strength, fatigue, insulin-resistance, higher rates of cardiovascular morbidity and reduced bone density. Exercise is an increasingly prescribed solution and it has been shown that cardiorespiratory fitness and physical activity have an important survival role but one that is often under-utilised. In terms of mortality, cardiovascular disease is the leading cause of death in patients with prostate cancer and exercise to increase physical activity is recommended in the American College of Sports Medicine's (ACSM) guidelines to counter this, given the clear cardioprotective effects it has.

The World Health Organisation defines the term "physical activity" as "any bodily movement produced by skeletal muscles that requires energy expenditure" and differentiates it from "exercise" which it defines as "a subcategory of physical activity that is planned, structured, repetitive, and purposeful" in order to improve or maintain physical fitness. There is good evidence from a systematic review and meta-analysis that exercise in patients with prostate cancer is safe, improves aerobic fitness and muscular strength, fatigue, body mass composition, quality of life and physical function.

There is no consensus over the detail of exercise prescription in cancer survivors and there are considerable differences between the protocols in studies to date. Many studies have employed moderate intensity activities such as cycling, jogging, walking or using a cross trainer but the frequency and duration employed have not been consistent, ranging from 2 to 7 days a week and 15-60 minutes per session.

Other than duration and frequency, one other important variable in exercise interventions is exercise intensity. The ACSM guidance highlights this as an area where knowledge is lacking and thus where further research is needed. In terms of physical activity in healthy populations, there is believed to be a dose-response relationship of volume with all-cause mortality, however, higher intensity might be able to produce similar results to increasing volume.

High intensity exercise is considered to be when a person exercises at greater than or equal to 80% of their maximal oxygen uptake capacity (VO2 MAX). In patients with cancer, intensity is the strongest component of an exercise regime that predicts improvements in quality of life. Higher intensity exercise can also lead to improvements in fatigue, aerobic fitness, muscle strength and function as well as an inverse link with the risk of premature death in cancer survivors.

The first interventions examining high intensity training in patients with prostate cancer employed sessions of 35 minutes with varying intervals from 1 - 25 minutes. These studies reported improvements in physiological function, such as reductions in fasting glucose and increases in the cardioprotective high-density lipoprotein. Subsequent studies have reproduced the physiological gains from high-intensity training and found them to be superior when compared to lower-intensity training. Even short interventions in cancer patients, such as 6 weeks, appear to provide significant improvements in VO2MAX.

Time and enjoyment are often cited barriers to regular physical activity and thus, high intensity interval training (HIIT) has been offered as a potential time-efficient solution that is perceived as more enjoyable than moderate continuous training in both healthy and cancer patients. HIIT can take a number of forms but a commonly employed protocol consists of 4-10 repeated maximal Wingate sprints with rest intervals in between. The total duration of the sessions, including the warm-up and warm-down, however, lasted a similar duration to the continuous moderate exertion aerobic exercise protocols. The protocol has, therefore, now been further condensed to reduced-exertion HIIT sessions (REHIT). This consists of 10 minutes of low intensity workload incorporating two or three 20 s Wingate sprints at set intervals. It was hypothesised by Metcalfe et al that, because energy stored in the muscle as glycogen was depleted to a similar extent in shorter 15-20 second sprints compared to the traditional 4-6 x 30 second sprints in HIIT, the shorter sprints would still produce physiological improvements. Indeed, REHIT improved both VO2MAX and insulin sensitivity.

Evidence that HIIT results in greater physiological benefits and for less time commitment than those achieved by continuous moderate intensity training in healthy populations is now well established and growing evidence replicates these findings in patients with cancer. REHIT could therefore provide patients with prostate cancer an opportunity to achieve at least the same physiological benefits as continuous moderate intensity training but with much less time commitment. The aim of this project is to investigate whether a REHIT intervention results in improved cardiorespiratory fitness in patients with prostate cancer.

Participants

For this pilot study, 30 patients who have been diagnosed with prostate cancer will be recruited from a number of Gloucestershire-based sites; a Macmillan Cancer Support initiative called Next Steps, a patient-let prostate cancer support group and the Gloucestershire Hospitals NHS Foundation Trust's uro-oncology specialist nurse service. Participants will be asked to give their written consent to participate in the study. Patients with activity status of "high", as assessed using the International Physical Activity Questionnaire (IPAQ), will be excluded from the study. The period of recruitment will be November 2017 to February 2019. Participants will be randomised to a control group or the exercise intervention group. The study will be subject to gaining ethical approval from the University of Bath Research Ethics Approval Committee and the NHS Research Ethics Committee.

Baseline Testing

The pre- and post-intervention cardiorespiratory fitness testing will be conducted at the University of Gloucestershire's Performance Laboratory. Pre-intervention maximal oxygen uptake capacity testing (VO2 max), will be performed at the initial visit to the laboratory. This will be determined using an incremental cycling test to volitional exhaustion on a cycle ergometer and a metabolic cart to analyse VO2 MAX. Patients will be asked to perform a 2-minute warm-up at 50 watts before an incremental 1 watt per 3 seconds to volitional exhaustion with verbal encouragement. VO2 MAX will be taken as the highest value in a 15-breath rolling average.

Experimental Procedures

Following baseline testing, participants in the exercise group will start a 6-week training protocol involving 3 sessions a week. The REHIT interventions will utilise a gym in Gloucestershire used by the Macmillan Cancer Support's Next Steps project. Each session will include 10 minutes of unloaded pedalling using a cycle ergometer. Volunteers will be asked to increase to their maximal pedal frequency possible for 1-2 seconds prior to applying a resistance of 5 % of pre-training body weight for the Wingate sprint. The sprints will take place at 2 minutes and at 6 minutes. Sprint duration will be increased from 10 seconds in the first week to 15 seconds in the second and third weeks and finally 20 seconds in the remaining weeks. Patients will receive strong verbal encouragement during the sprints after which the resistance will be removed. The acceptability of the training will be assessed with a questionnaire based on that used by Boereboom et al. in 2016. Participants in the control group will be asked to continue with their usual care and lifestyle activities.

Statistical Analysis

Data will be presented as mean ± standard deviation. Statistical analysis will be performed using SPSS statistical software. Paired sample T-tests will be used to analyse differences in pre- and post-intervention VO2MAX. Statistical significance will be accepted at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* For this pilot study, we will aim to recruit a total of 30 patients who have been diagnosed with prostate cancer. They will be recruited from a number of Gloucestershire-based sites; a Macmillan Cancer Support initiative called Next Steps, a patient-let prostate cancer support group and the Gloucestershire Hospitals NHS Foundation Trust's uro-oncology specialist nurse service. Participants will be asked to give their written consent to participate in the study. All participants will be given written and verbal information on what the study involves and will be able to ask any questions they may have. The subjects will all be informed that they may withdraw from the study at any point, without giving a reason.

Exclusion Criteria:

* Any cardiovascular condition with the exception of well-controlled uncomplicated hypertension treated with no more than two drugs (either an ACE, ARB, calcium channel blocker, or diuretic)
* Cerebrovascular disease including previous stroke or aneurysm
* History of exercise-induced asthma
* Any prior history of malignancy with the exception of basal cell carcinoma of the skin
* BMI>35 kg/m¬2
* Uncontrolled hypertension (systolic blood pressure >160 mm Hg and/or diastolic blood pressure >100 mm Hg after at least a 5 minute seated rest at the screening visit)
* A clinically significant ECG abnormality at the screening visit which in the opinion of the investigators exposes the subject to risk by enrolling in the trial
* Overt contraindications to exercise as determined with a normal resting ECG
* 'Yes' to any questions on a standard physical activity readiness questionnaire (PAR¬Q)
* Classification as highly physically active on the International Physical Activity Questionnaire (IPAQ)
* Inability to fully understand the verbal and written descriptions of the study in English, and the instructions provided during the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only patients with prostate cancer will be eligible and therefore this study will only include male patients.
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Change from baseline Pre- and post- 6-week exercise intervention
  Cardiorespiratory fitness using maximal oxygen uptake capacity testing (VO2 max)

SECONDARY OUTCOMES:
Peripheral blood pressure | Change from baseline Pre- and post- 6-week exercise intervention
  Peripheral blood pressure using a sphygmomanometer
Central blood pressure and arterial stiffness | Change from baseline Pre- and post- 6-week exercise intervention
  Central blood pressure will be assessd using pulse wave analysis, a non-invasive assessment described by Wang et al. (2010) using two blood pressure cuffs situated over the brachial and femoral arteries, and a tonometer. Carotid artery stiffness and velocity will be assessed using Doppler ultrasound
Arterial stiffness | Change from baseline Pre- and post- 6-week exercise intervention
  Carotid artery stiffness and velocity will be assessed using Doppler ultrasound
Tissue saturation index of vastus lateralis and rectus femoris | Change from baseline Pre- and post- 6-week exercise intervention
  Tissue saturation index of vastus lateralis and rectus femoris muscles will be assessed using continuous wave near infrared spectroscopy.
Height | Change from baseline Pre- and post- 6-week exercise intervention
  Measured in metres and then aggregated with weight in kilograms to produce BMI in kg/m^2
Weight | Change from baseline Pre- and post- 6-week exercise intervention
  Measured in kilograms and then aggregated with height in metres to produce BMI in kg/m^2
Quality of life measure | Change from baseline Pre- and post- 6-week exercise intervention
  Quality of life measure using SF-36®
Body composition | Change from baseline Pre- and post- 6-week exercise intervention
  Body composition using air displacement plethysmography in a Cosmed Bod Pod®.
Reduced-exertion high intensity interval training acceptability questionnaire | Immediately post-6 week exercise intervention
  The acceptability of the training will be assessed with a questionnaire based on that used by (Boereboom et al., 2016).

CONTACTS AND LOCATIONS:
Overall Officials: James Turner, PhD, Principal Investigator — University of Bath
Locations (1):
- Gloucestershire Care Services NHS Trust, Gloucester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adamsen L, Quist M, Andersen C, Moller T, Herrstedt J, Kronborg D, Baadsgaard MT, Vistisen K, Midtgaard J, Christiansen B, Stage M, Kronborg MT, Rorth M. Effect of a multimodal high intensity exercise intervention in cancer patients undergoing chemotherapy: randomised controlled trial. BMJ. 2009 Oct 13;339:b3410. doi: 10.1136/bmj.b3410. PMID 19826172
- [Background] Bartlett JD, Close GL, MacLaren DP, Gregson W, Drust B, Morton JP. High-intensity interval running is perceived to be more enjoyable than moderate-intensity continuous exercise: implications for exercise adherence. J Sports Sci. 2011 Mar;29(6):547-53. doi: 10.1080/02640414.2010.545427. PMID 21360405
- [Background] Boereboom CL, Phillips BE, Williams JP, Lund JN. A 31-day time to surgery compliant exercise training programme improves aerobic health in the elderly. Tech Coloproctol. 2016 Jun;20(6):375-382. doi: 10.1007/s10151-016-1455-1. Epub 2016 Mar 25. PMID 27015678
- [Background] Bourke L, Smith D, Steed L, Hooper R, Carter A, Catto J, Albertsen PC, Tombal B, Payne HA, Rosario DJ. Exercise for Men with Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol. 2016 Apr;69(4):693-703. doi: 10.1016/j.eururo.2015.10.047. Epub 2015 Nov 26. PMID 26632144
- [Background] Buchheit M, Laursen PB. High-intensity interval training, solutions to the programming puzzle. Part II: anaerobic energy, neuromuscular load and practical applications. Sports Med. 2013 Oct;43(10):927-54. doi: 10.1007/s40279-013-0066-5. PMID 23832851
- [Background] Despres JP. Physical Activity, Sedentary Behaviours, and Cardiovascular Health: When Will Cardiorespiratory Fitness Become a Vital Sign? Can J Cardiol. 2016 Apr;32(4):505-13. doi: 10.1016/j.cjca.2015.12.006. Epub 2015 Dec 15. PMID 26907579
- [Background] Devin JL, Sax AT, Hughes GI, Jenkins DG, Aitken JF, Chambers SK, Dunn JC, Bolam KA, Skinner TL. The influence of high-intensity compared with moderate-intensity exercise training on cardiorespiratory fitness and body composition in colorectal cancer survivors: a randomised controlled trial. J Cancer Surviv. 2016 Jun;10(3):467-79. doi: 10.1007/s11764-015-0490-7. Epub 2015 Oct 19. PMID 26482384
- [Background] Ferrer RA, Huedo-Medina TB, Johnson BT, Ryan S, Pescatello LS. Exercise interventions for cancer survivors: a meta-analysis of quality of life outcomes. Ann Behav Med. 2011 Feb;41(1):32-47. doi: 10.1007/s12160-010-9225-1. PMID 20931309
- [Background] Gibala MJ, Little JP, Macdonald MJ, Hawley JA. Physiological adaptations to low-volume, high-intensity interval training in health and disease. J Physiol. 2012 Mar 1;590(5):1077-84. doi: 10.1113/jphysiol.2011.224725. Epub 2012 Jan 30. PMID 22289907
- [Background] Gillen JB, Gibala MJ. Is high-intensity interval training a time-efficient exercise strategy to improve health and fitness? Appl Physiol Nutr Metab. 2014 Mar;39(3):409-12. doi: 10.1139/apnm-2013-0187. Epub 2013 Sep 27. PMID 24552392
- [Background] Hamer M, Stamatakis E, Saxton JM. The impact of physical activity on all-cause mortality in men and women after a cancer diagnosis. Cancer Causes Control. 2009 Mar;20(2):225-31. doi: 10.1007/s10552-008-9237-3. Epub 2008 Oct 2. PMID 18830799
- [Background] Hvid T, Winding K, Rinnov A, Dejgaard T, Thomsen C, Iversen P, Brasso K, Mikines KJ, van Hall G, Lindegaard B, Solomon TP, Pedersen BK. Endurance training improves insulin sensitivity and body composition in prostate cancer patients treated with androgen deprivation therapy. Endocr Relat Cancer. 2013 Aug 19;20(5):621-32. doi: 10.1530/ERC-12-0393. Print 2013 Oct. PMID 23744766
- [Background] Lakoski SG, Willis BL, Barlow CE, Leonard D, Gao A, Radford NB, Farrell SW, Douglas PS, Berry JD, DeFina LF, Jones LW. Midlife Cardiorespiratory Fitness, Incident Cancer, and Survival After Cancer in Men: The Cooper Center Longitudinal Study. JAMA Oncol. 2015 May;1(2):231-7. doi: 10.1001/jamaoncol.2015.0226. PMID 26181028
- [Background] Laukkanen JA, Rauramaa R, Makikallio TH, Toriola AT, Kurl S. Intensity of leisure-time physical activity and cancer mortality in men. Br J Sports Med. 2011 Feb;45(2):125-9. doi: 10.1136/bjsm.2008.056713. Epub 2009 Jul 28. PMID 19656766
- [Background] Mann T, Lamberts RP, Lambert MI. Methods of prescribing relative exercise intensity: physiological and practical considerations. Sports Med. 2013 Jul;43(7):613-25. doi: 10.1007/s40279-013-0045-x. PMID 23620244
- [Background] Martin E, Battaglini C, Hands B, Naumann FL. Higher-intensity exercise helps cancer survivors remain motivated. J Cancer Surviv. 2016 Jun;10(3):524-33. doi: 10.1007/s11764-015-0498-z. Epub 2015 Nov 19. PMID 26586495
- [Background] Martin EA, Battaglini CL, Hands B, Naumann F. Higher-Intensity Exercise Results in More Sustainable Improvements for VO2peak for Breast and Prostate Cancer Survivors. Oncol Nurs Forum. 2015 May;42(3):241-9. doi: 10.1188/15.ONF.42-03AP. PMID 25901376
- [Background] Metcalfe RS, Babraj JA, Fawkner SG, Vollaard NB. Towards the minimal amount of exercise for improving metabolic health: beneficial effects of reduced-exertion high-intensity interval training. Eur J Appl Physiol. 2012 Jul;112(7):2767-75. doi: 10.1007/s00421-011-2254-z. Epub 2011 Nov 29. PMID 22124524
- [Background] Metcalfe RS, Koumanov F, Ruffino JS, Stokes KA, Holman GD, Thompson D, Vollaard NB. Physiological and molecular responses to an acute bout of reduced-exertion high-intensity interval training (REHIT). Eur J Appl Physiol. 2015 Nov;115(11):2321-34. doi: 10.1007/s00421-015-3217-6. Epub 2015 Jul 9. PMID 26156806
- [Background] Nguyen PL, Alibhai SM, Basaria S, D'Amico AV, Kantoff PW, Keating NL, Penson DF, Rosario DJ, Tombal B, Smith MR. Adverse effects of androgen deprivation therapy and strategies to mitigate them. Eur Urol. 2015 May;67(5):825-36. doi: 10.1016/j.eururo.2014.07.010. Epub 2014 Aug 2. PMID 25097095
- [Background] Quist M, Rorth M, Zacho M, Andersen C, Moeller T, Midtgaard J, Adamsen L. High-intensity resistance and cardiovascular training improve physical capacity in cancer patients undergoing chemotherapy. Scand J Med Sci Sports. 2006 Oct;16(5):349-57. doi: 10.1111/j.1600-0838.2005.00503.x. PMID 16978255
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Soerjomataram I, Lortet-Tieulent J, Parkin DM, Ferlay J, Mathers C, Forman D, Bray F. Global burden of cancer in 2008: a systematic analysis of disability-adjusted life-years in 12 world regions. Lancet. 2012 Nov 24;380(9856):1840-50. doi: 10.1016/S0140-6736(12)60919-2. Epub 2012 Oct 16. PMID 23079588
- [Background] Toohey K, Pumpa KL, Arnolda L, Cooke J, Yip D, Craft PS, Semple S. A pilot study examining the effects of low-volume high-intensity interval training and continuous low to moderate intensity training on quality of life, functional capacity and cardiovascular risk factors in cancer survivors. PeerJ. 2016 Oct 20;4:e2613. doi: 10.7717/peerj.2613. eCollection 2016. PMID 27781180
- [Background] Wang KL, Cheng HM, Sung SH, Chuang SY, Li CH, Spurgeon HA, Ting CT, Najjar SS, Lakatta EG, Yin FC, Chou P, Chen CH. Wave reflection and arterial stiffness in the prediction of 15-year all-cause and cardiovascular mortalities: a community-based study. Hypertension. 2010 Mar;55(3):799-805. doi: 10.1161/HYPERTENSIONAHA.109.139964. Epub 2010 Jan 11. PMID 20065155
- [Background] Ware, J.E., Snow, K.K., Kosinski, M., Gandek, B. SF-36® Health Survey Manual and Interpretation Guide. Boston, MA: New England Medical Center, The Health Institute, 1993
- [Background] Weston M, Taylor KL, Batterham AM, Hopkins WG. Effects of low-volume high-intensity interval training (HIT) on fitness in adults: a meta-analysis of controlled and non-controlled trials. Sports Med. 2014 Jul;44(7):1005-17. doi: 10.1007/s40279-014-0180-z. PMID 24743927
- [Background] Global Recommendations on Physical Activity for Health. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK305057/ PMID 26180873